CLINICAL TRIAL: NCT06153082
Title: Rotational Thromboelastometry [ROTEM] vs Thromboelastography [TEG] Guided Blood Component Use in Patients With Cirrhosis of Liver With Nonvariceal Bleeding: A Randomized Controlled Trial
Brief Title: Rotational Thromboelastometry [ROTEM] vs Thromboelastography [TEG] Guided Blood Component Use in Patients With Cirrhosis of Liver With Non-variceal Bleeding.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-69
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Thrombelastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROTEM Group (Experimental): In ROTEM group if CT EXTEM >80S FFP at dose of 10ml/kg or PCC 20-25IU/kg ,if MCF EXTEM <35 and MCF FIBTEM <8 CRYO or Fibrinogen concentrate, if MCF EXTEM<35 and MCF FIBTEM >8 Platelet, CL LY>50 Trenaxemic acid.
  Interventions: Diagnostic Test: ROTEM
- THROMBOELASTOGRAPHY (Active Comparator): Patients in the TEG group received blood components using the following triggers: FFP at a dose of 10 mL/kg of ideal body weight when reaction time (R time) was greater than 10 minutes; a single-donor apheresis platelet (SDAP) unit, which corresponds to approximately 6 to 8 pooled units of PLTs, transfused when the maximum amplitude (MA) was less than 55 mm; and cryoprecipitate (5 pooled units) transfused when the alpha angle was less than 45°
  Interventions: Diagnostic Test: Thromboelastography

INTERVENTIONS:
Diagnostic Test: ROTEM — In ROTEM group if CT EXTEM >80S FFP at dose of 10ml/kg or PCC 20-25IU/kg ,if MCF EXTEM <35 and MCF FIBTEM <8 CRYO or Fibrinogen concentrate, if MCF EXTEM<35 and MCF FIBTEM >8 Platelet, CL LY>50 Trenaxemic acid
  Arms: ROTEM Group
Diagnostic Test: Thromboelastography — Patients in the TEG group received blood components using the following triggers: FFP at a dose of 10 mL/kg of ideal body weight when reaction time (R time) was greater than 10 minutes; a single-donor apheresis platelet (SDAP) unit, which corresponds to approximately 6 to 8 pooled units of PLTs, transfused when the maximum amplitude (MA) was less than 55 mm; and cryoprecipitate (5 pooled units) transfused when the alpha angle was less than 45°.
  Arms: THROMBOELASTOGRAPHY

SUMMARY:
This study is aim to compare ROTEM and TEG guided coagulopathy correction in cirrhosis with non- variceal bleed.There are no other study in literature to compare this two group in cirrhosis with non-variceal bleed.This study will also assess the volume of blood product transfused with this two groups and it will compare among two groups.This will lessen the blood product transfusion and risk of transfusion relatedated complication.

DETAILED DESCRIPTION:
AIM:- To compare Rotational thrombo- elastometry vs Thrombo- elastography as a guide for blood component transfusion in patients of Cirrhosis with nonvariceal bleeding.

Methodology:- After fulfilling all inclusion and exclusion criteria, patients were randomized to either the TEG or ROTEM group in a 1:1 proportion. Patients in the TEG group received blood components using the following triggers: FFP at a dose of 10 mL/kg of ideal body weight when reaction time (R time) was greater than 10 minutes; a single-donor apheresis platelet (SDAP) unit, which corresponds to approximately 6 to 8 pooled units of PLTs, transfused when the maximum amplitude (MA) was less than 55 mm; and cryoprecipitate (5 pooled units) transfused when the alpha angle was less than 45°.In ROTEM group if CT EXTEM >80S FFP at dose of 10ml/kg or PCC 20-25IU/kg ,if MCF EXTEM <35 and MCF FIBTEM <8 CRYO or Fibrinogen concentrate, if MCF EXTEM<35 and MCF FIBTEM >8 Platelet, CL LY>50 Trenaxemic acid

Study population: patients with Cirrhosis of liver with nonvariceal bleeding Study design: Randomized controlled trial Study period: 1 years after ethical clearance

Sample size: Assuming that total volume of FFP used in TEG 760 ± 370 and further in ROTEM volume used 510±275 with α 5% power 90, we need to enrol 72 cases. Further assuming 10% inadequacy We had decided to enroll a total of 80 patients, 40 in each group.The allocation will be done randomly by block randomization method.

Monitoring and assessment: All the parameters of the objective and also noted any adverse effects.

STATISTICAL ANALYSIS:

The data will be entered in Microsoft excel and will be analyzed using SPSS version 22. The categorical data will be analyzed using Chi square/Fissure test. Exact test and continuous data will be compiled using t-test. Besides this the univariate and multivariate survival analysis will be carried out using Cox regression method. Kaplan-Meier technique will be applied for further analysis. P-value<0.05 will be considered as significant.

Adverse effects:Transfusion related complication

Stopping rule: If patient decided to withdraw from study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Cirrhosis of any etiology
2. Age between 18 and 80 years;
3. Presenting with nonvariceal upper GI bleeding (diagnosed after doing upper GI endoscopy, which showed ongoing
4. bleed form a nonvariceal source); and
5. Significant coagulopathy assessed by CCTs (INR > 1.8 and/or PLTs < 50 × 109/L).

Exclusion Criteria:

1. Variceal bleed
2. Post Variceal ligation ulcer bleed
3. Previous or current thrombotic events defined as any documented blood clot in a venous or arterial vessel;
4. Anti-PLT or anticoagulant therapy at the time of enrollment or that had been discontinued less than 7 days before evaluation for the study;
5. Pregnancy
6. Significant cardiopulmonary diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative volume of FFP transfused at Day 5. | Day 5

SECONDARY OUTCOMES:
Cumulative volume of Cryoprecipitate in both groups | 6 weeks
Cumulative volume of Platelet in both groups | 6 weeks
Cumulative volume of Trenaxemic acid Transfusion related reactions in both groups | 6 weeks
Duration of intensive care unit (ICU) in both groups | 6 weeks
Duration of hospital stay in both groups | 6 weeks
Survival in both groups at 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Saurav Paul, New Delhi, National Capital Territory of Delhi, India